CLINICAL TRIAL: NCT01780272
Title: A Trial to Investigate the Impact of Nocturnal Hypoglycaemia on Sleep in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: NN1250-3997; U1111-1127-4819 (Other: WHO)
Record Dates: First submitted 2013-01-17; First posted 2013-01-31 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normoglycaemia followed by hypoglycaemia (Other)
  Interventions: Other: glucose clamp
- Hypoglycaemia followed by normoglycaemia (Other)
  Interventions: Other: glucose clamp

INTERVENTIONS:
Other: glucose clamp — Each subject will complete one adaptation night visit followed by two experimental night visits, one normoglycaemic and one hypoglycaemic, in randomised order. While subjects are asleep, sleep patterns will be monitored online using polysomnographic recordings during a hypoglycaemic and a normoglycaemic clamp (using constant intravenous (i.v.) infusion of human soluble insulin (Actrapid®)). Plasma glucose will be monitored.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the impact of low blood sugar during the night on sleep in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 24 weeks prior to screening
* Currently treated with any anti-diabetic treatment (incl. diet and exercise) except insulin with a stable dose for more than 4 weeks prior to screening
* Body mass index below 35 kg/m^2

Exclusion Criteria:

* Severe hypoglycaemic event during the past 6 months or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Any other chronic disorder or severe disease by clinical information (including chronic obstructive pulmonary disease (COPD), sleep apnoea and epilepsy) which, in the opinion of the investigator might jeopardise subject's sleep, safety or compliance with the protocol, or subjects with mental incapacity or language barriers precluding adequate understanding or co-operation or who, in the opinion of the investigator, should not participate in the trial
* Use of antidepressants, antipsychotics, hypnotics, sedatives or other drugs known to influence sleep within 12 weeks prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The number of electroencephalogram (EEG) identified arousals | During the first four hours (0-4 hours) after reaching sleep stage N2

SECONDARY OUTCOMES:
Time spent in the different sleep stages (% of total sleep time): Sleep stage N1, Sleep stage N2, Sleep stage N3 and Rapid Eye Movement (REM) sleep | During the first four hours (0-4 hours) after reaching sleep stage N2
Total sleep time | 0-8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Glostrup Municipality, Denmark

REFERENCES:
- [Result] Jennum P, Stender-Petersen K, Rabol R, Jorgensen NR, Chu PL, Madsbad S. The Impact of Nocturnal Hypoglycemia on Sleep in Subjects With Type 2 Diabetes. Diabetes Care. 2015 Nov;38(11):2151-7. doi: 10.2337/dc15-0907. Epub 2015 Sep 25. PMID 26407587
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com